CLINICAL TRIAL: NCT05929235
Title: A Phase 1, First-in-Human, Dose-Escalation and Expansion Study of FX-909 (as Monotherapy or in Combination With Pembrolizumab) in Patients With Advanced Solid Malignancies, Including Advanced Urothelial Carcinoma
Brief Title: A Study of FX-909 in Patients With Advanced Solid Malignancies, Including Advanced Urothelial Carcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Flare Therapeutics Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FX-909-CLINPRO-1; 3. KEYNOTE-G54 4. MK-3475-G54 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2023-05-30; First posted 2023-07-03 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Advanced Urothelial Carcinoma; Oral Drug Administration; Open Label
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Part A is a 3+3 dose escalation design. Part B will proceed in a 2-stage design that will investigate 2 dose arms of FX-909 in Stage 1; with a single arm in Stage 2 envisioned. Part 1A1 is a dose escalation to investigate FX-909 in combination with Pembrolizumab.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Escalation (Experimental): 3+3 design, 5 dose levels
  Interventions: Drug: FX-909
- Expansion Expansion (Experimental): Part B will proceed in a 2-stage design that will investigate 2 dose arms of FX-909 in Stage 1; with a single arm in Stage 2 envisioned.
  Interventions: Drug: FX-909
- FX-909 in Combination with Pembrolizumab (Experimental): Part 1A1 will be a dose-escalation study to investigate FX-909 in combination with Pembrolizumab.
  Interventions: Drug: FX-909; Drug: Pembrolizumab (KEYTRUDA ®); Drug: KEYTRUDA ®( Pembrolizumab)

INTERVENTIONS:
Drug: FX-909 — FX-909 is an orally available new molecular entity that inhibits basal- and ligand-activated transcription by PPARG.
Drug: Pembrolizumab (KEYTRUDA ®) — Pembrolizumab is an immunotherapy checkpoint inhibitor.
  Arms: FX-909 in Combination with Pembrolizumab
Drug: KEYTRUDA ®( Pembrolizumab) — Keytruda is an immunotherapy checkpoint inhibitor.
  Arms: FX-909 in Combination with Pembrolizumab

SUMMARY:
The goal of this clinical trial is to study the safety and tolerability in all advanced solid tumors, including advanced urothelial carcinoma.

The main question[s] it aims to answer are:

* Is FX-909 safe and tolerable, as a monotherapy and in combination with Pembrolizumab
* What is the right dose level for patients

Participants will be asked to take FX-909 daily in tablet form, or FX-909 daily and Pembrolizumab every 3 weeks, and record any outcomes from taking the drug. Participants will also be asked to return for multiple site visits for various blood tests and to collect blood and tumor samples as well as have regular CT/MRI scans.

DETAILED DESCRIPTION:
This is an open-label Phase 1 study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary clinical activity of FX-909 given orally (PO) in patients with advanced solid malignancies. Initially, FX-909 will be given in a dose-escalation phase (Part A) to determine the preliminary recommended phase 2 dose (RP2D). Part B will be a dose expansion phase to further evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and clinical activity of FX-909 in patients with locally advanced (unresectable) and metastatic urothelial carcinoma. Part 1A1 will be a dose escalation of FX-909 in combination with Pembrolizumab. Throughout the study patients will be treated in 28 or 21-day cycles.

ELIGIBILITY:
Part A/B Inclusion Criteria:

1. Able to understand and willing to sign an informed consent.
2. Age ≥ 18 years.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2.
4. An archival, paraffin-embedded, formalin-fixed, tumor sample (see Laboratory Manual for details) that in Part A is no more than 30 months old at the time of screening or in Part B is no more than 30 months old at time of pre-screening. If an archival tumor sample is not available or is older than 30 months, then the patient must consent to provide a fresh biopsy during screening.
5. Part A: Histologically or cytologically diagnosed, locally advanced (unresectable) or metastatic solid malignancies that have progressed after all available standard therapy for the specific tumor type, or for which no standard therapy exists. Patients for whom standard therapies are intolerable or considered inappropriate by the Investigator are eligible.

   Part B: Patients with histologically or cytologically confirmed, locally advanced (unresectable) or metastatic urothelial carcinoma exhibiting high levels of PPARG protein expression will be prospectively enrolled in this study. Eligibility will require a Tumor Positivity Score (TPS) of ≥ 60%, as determined by an investigational immunohistochemistry (IHC) assay for PPARG.

   • Treated with ≤ 4 prior therapies for advanced or metastatic disease Patients in Part B must have progressed after all available standard therapy, been unable to tolerate standard therapy, or be considered inappropriate for standard therapy by the Investigator.
6. Part A: Patients with or without measurable disease (as defined by RECIST version 1.1) will be eligible for enrollment.

Part B: Patients must have measurable disease per RECIST version 1.1 with ≥ 1 site of measurable disease that has not been previously irradiated or has progressed after radiation therapy.

7. Screening laboratory values meet the criteria outlined in Table 8.

o Hematologic criteria may be met with transfusion of blood products or administration of G-CSF, provided they are not given within 7 days prior to enrollment. Hematologic parameters must meet the inclusion criteria prior to dosing on Cycle 1 Day 1.

Part A/B Exclusion Criteria:

1. Female patients who are pregnant (confirmed with a positive pregnancy test) or breastfeeding.
2. Prior anticancer chemotherapy or small molecule targeted therapy, either investigational or commercially approved and available, within 2 weeks or 5 half-lives (whichever is shorter) prior to the start of study drug administration. When the most recent therapy was a biological therapy (including antibody-drug conjugates), an immune-checkpoint inhibitor (eg, anti-PD(L)1 or anti-CTLA4), or immune agonist, patients should wait 4 weeks before starting therapy with FX-909. (See Exclusion Criterion 6 for required radiotherapy windows.)
3. Prior therapy directly inhibiting PPARG or RXRA.
4. Adverse events from prior therapy that have not returned to baseline or stabilized at Grade 1 (except alopecia, hearing loss, vitiligo, endocrinopathy managed with replacement therapy, and Grade ≤ 2 neuropathy) prior to study drug administration.
5. Prior major surgery (excluding placement of vascular access) within 4 weeks before study drug administration.
6. Prior radiation therapy with an inadequate washout between the last dose and the start of study drug, defined as follows: 1) at least 2 weeks for palliative radiation to the extremities for osseous bone metastases is required; and 2) at least 4 weeks for radiation to non-extremity sites is required.
7. History of another malignancy in the previous 2 years, unless cured by surgery alone and continuously disease free. Exceptions include appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, melanoma in situ status-post full-thickness resection without recurrence, Stage 1 uterine cancer, localized prostate cancer that has been treated surgically with curative intent and presumed cured, or other malignancies with an expected curative outcome. Patients requiring adjuvant therapy within the past 2 years for another malignancy will not be considered to have been cured.
8. QT interval corrected using Fridericia's Formula (QTcF) >470 msec in screening, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in first degree relatives.
9. Known active diagnosis of lipodystrophy/lipoatrophy, or an ongoing need to receive medications known to cause lipodystrophy/lipoatrophy.
10. Any active uncontrolled systemic bacterial, viral, or fungal infection requiring treatment.
11. Known history of HIV seropositivity. Those who have no detectable viral load on highly active antiretroviral therapy (HAART) are permitted.
12. Patients with chronic hepatitis B virus (HBV) infection. Patients are permitted with either universal prophylaxis or a pre-emptive treatment approach consistent with regional or national guidelines for patients who receive anticancer therapies.
13. Active hepatitis C virus (HCV) infection. Those who have completed curative therapy for HCV and have no detectable viral load are permitted.
14. Prior diagnosis of chronic or recurrent (> 1 episode) pancreatitis at any time or a diagnosis of acute pancreatitis within the 6 months prior to screening.
15. Significant impairment of lung function indicated by resting oxygen saturations below 92% on room air or requiring chronic use of ambulatory supplemental oxygen.
16. Uncontrolled or symptomatic central nervous system (CNS) metastases, leptomeningeal disease, or carcinomatous meningitis. Asymptomatic brain metastasis is allowed if they have been stable after appropriate radiotherapy for 1 month.
17. Need for treatment with high doses of oral or intravenous steroids (> 10 mg/day prednisone or equivalent). Physiologic doses of corticosteroids for treatment of endocrinopathies may be continued if the patient is on a stable dose for at least 1 month.
18. Need or anticipated need for treatment with a prohibited therapy during the treatment phase of this study.
19. Concurrent participation in any other investigational therapeutic study.
20. History of any of the following cardiovascular diseases:

    o Recent history (within the 6 months prior to screening) of serious uncontrolled cardiac arrhythmia (including atrial fibrillation without adequate rate control) or clinically significant ECG abnormalities including second-degree (Type II) or third-degree atrioventricular node block

    o Documented cerebrovascular event (stroke or transient ischemic attack), cardiomyopathy, myocardial infarction, acute coronary syndromes (including unstable angina pectoris), coronary angioplasty, stenting, or bypass grafting within the 6 months prior to enrollment
    * Congestive heart failure (Class III or IV) as defined by the New York Heart Association functional classification system
    * Recent history (within the past 6 months) of symptomatic pericarditis
21. Thromboembolic events and/or bleeding disorders ≤ 28 days (eg, deep vein thrombosis or pulmonary embolism) prior to the first dose of study drug.
22. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which, in the Investigator's opinion, makes it undesirable for the patient to participate in the study or would jeopardize compliance with the protocol.
23. Patients with type 1 diabetes mellitus, or type 2 diabetes mellitus that is not adequately controlled with diet, exercise, or oral hypoglycemic agents and/or injectable agents other than insulin (as defined by HbA1c and fasting plasma glucose criteria in Table 8. Patients taking insulin are excluded from the study. Medication for type 2 diabetes mellitus should have remained stable for the past 14 days prior to screening).
24. Known hypersensitivity to FX-909 or any of its excipients.
25. Patients with gastrointestinal disorders that may interfere with the ability to swallow tablets or absorb study medication.
26. Patient is or has an immediate family member (eg, spouse, parent/legal guardian, sibling, or child) who is a member of the study site or Sponsor staff directly involved with this study, unless prospective Institutional Review Board (IRB) or Ethics Committee (EC) approval (by chair or designee) is given allowing exception to this criterion for a specific patient.
27. Patients with any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before study entry.
28. Any condition that, in the opinion of the Investigator, would interfere with evaluation of the investigational product or interpretation of the patient's safety or study results.

Part 1A1 Inclusion Criteria:

1. Able to understand and willing to sign an informed consent 2. Aged 18 years or older on the day written informed consent is given 3. ECOG performance status 0 or 1 4. Histologically or cytologically confirmed, locally advanced (unresectable) or metastatic urothelial carcinoma by pathology report.

5. Participants must have received and progressed after all available standard therapies known to confer clinical benefit, been unable to tolerate standard therapy, or be considered inappropriate for standard therapy by the Investigator.

6. Must have progressed on treatment with an anti-PD-1/L1 mAb administered either as monotherapy or in combination with other checkpoint inhibitors or other therapies. PD-1 treatment progression is defined by meeting all of the following criteria:

1. Received at least 2 doses of an approved anti-PD-1/L1 mAb.
2. Documented disease progression after anti-PD-1/L1 treatment (consistent with the principles of RECIST v1.1). The initial evidence of disease progression is to be confirmed by a second assessment no less than 4 weeks from the date of the first documented disease progression, in the absence of rapid clinical progression (as defined in 2.c).
3. Progressive disease has been documented within 12 weeks from the last dose of anti-PD-1/L1 mAb.

   1. Progressive disease is determined consistent with the principles of RECIST v1.1.
   2. This determination is made by the investigator. Once disease progression is confirmed, the initial date of disease progression documentation will be considered the date of disease progression.

   7. Measurable disease per RECIST 1.1 as assessed by the local site investigator/radiology. Lesions situated in a previously irradiated area are considered measurable if progression has been shown in such lesions.

   8. Archival tumor tissue sample within 30 months of enrollment or newly obtained [core, incisional, OR excisional] biopsy of a tumor lesion not previously irradiated has been provided.

   9. Participants who have AEs due to previous anticancer therapies (with the exception of alopecia or peripheral sensory neuropathy) must have recovered to ≤Grade 1 or baseline. Participants with endocrine-related AEs who are adequately treated with hormone replacement are eligible, as are participants with ≤Grade 2 neuropathy, hearing loss, or alopecia.

   10. If male, agrees to use an adequate method of contraception starting with the first dose of study drug through 90 days after the last dose of study drug. Please see Section 10.3 for a list of acceptable birth control methods. Male participants must not donate sperm throughout the study period and for 90 days after the last dose of the study treatment.

   11. Female participants of childbearing potential must have a negative serum pregnancy test at screening within 7 days of the Cycle 1 Day 1 dosing. Female participants of childbearing potential must agree to use a highly effective form of contraception, as defined in the protocol (Section 10.3), during the study and for 120 days after the last dose of study drug. To be considered NOT of childbearing potential, female participants must have had a hysterectomy or bilateral oophorectomy or be 1-year post-menopause or have had amenorrhea for a period of 12 months or longer in the absence of chemotherapy, anti-estrogens, or ovarian suppression.

   12. HIV-infected participants must have well controlled HIV on ART, defined as:

<!-- -->

1. Participants on ART must have a CD4+ T-cell count ≥350 cells/mm3 at the time of screening
2. Participants on ART must have achieved and maintained virologic suppression, defined as confirmed HIV RNA level below 50 or the LLOQ (below the limit of detection) using the locally available assay at the time of screening and for at least 12 weeks before screening
3. It is advised that participants must not have had any AIDS-defining opportunistic infections within the past 12 months
4. Participants on ART must have been on a stable regimen, without changes in drugs or dose modification, for at least 4 weeks before study entry (Day 1) and agree to continue ART throughout the study.
5. Participants with HIV should continue ongoing management by their health care provider(s), including monitoring of HIV viral load, CD4+ T-cell count, and appropriate supportive care measures.

   13. Participants who are HBsAg positive are eligible if they have received HBV antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to randomization.

a. Hepatitis B screening tests are not required unless:

1. Known history of HBV infection
2. As mandated by local guidelines

14. Participants with a history of HCV infection are eligible if HCV viral load is undetectable at screening.

Note: Participants must have completed curative antiviral therapy at least 4 weeks prior to randomization.

1. Hepatitis C screening tests are not required unless:

   3. Known history of HCV infection 4. As mandated by local guidelines 15. Adequate organ function as defined in Table 20.

Part 1A1 Exclusion Criteria:

1. HIV-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease.
2. Participants with type 1 diabetes mellitus, or type 2 diabetes mellitus that is not adequately controlled with diet, exercise, or oral hypoglycemic agents and/or injectable agents other than insulin (as defined by HbA1c and fasting plasma glucose criteria in Table 20. Participants taking insulin are excluded from the study. Medication for type 2 diabetes mellitus should have remained stable for the past 14 days prior to screening).
3. Participants with gastrointestinal disorders that may interfere with the ability to swallow tablets or absorb study medication.
4. Thromboembolic events and/or bleeding disorders ≤28 days (eg, deep vein thrombosis or pulmonary embolism) prior to the first dose of study drug.

   Prior/Concomitant Therapy
5. Prior therapy inhibiting PPARG or RXRA.
6. Received any prior immunotherapy and was discontinued from that treatment due to a Grade 3 or higher irAE (except endocrine disorders that can be treated with replacement therapy) or was discontinued from that treatment due to Grade 2 myocarditis or recurrent Grade 2 pneumonitis.
7. Received prior systemic anticancer therapy within 2 weeks or 5 half-lives (whichever is shorter) before the start of study drug administration. When the most recent therapy was a biological therapy (including antibody-drug conjugates), an immune-checkpoint inhibitor (eg, anti-PD(L)1 or anti-CTLA4), or immune agonist, participants should wait 4 weeks before starting therapy with FX-909.
8. Note: If participant underwent major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
9. Received prior radiotherapy within 2 weeks of the start of study intervention, or has radiation-related toxicities, requiring corticosteroids.
10. Note: Two weeks or fewer of palliative radiotherapy for non-CNS disease is permitted. The last radiotherapy treatment must have been performed at least 7 days before the first dose of study intervention.
11. Received a live or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed.

    Prior/Concurrent Clinical Study Experience
12. Has received an investigational agent or has used an investigational device within 4 weeks prior to study intervention administration.

    Diagnostic Assessments
13. Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in doses exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study intervention.
14. Prior diagnosis of chronic or recurrent (> 1 episode) pancreatitis at any time or a diagnosis of acute pancreatitis within the 6 months prior to screening,
15. Significant impairment of lung function indicated by resting oxygen saturations below 92% or requiring chronic use of ambulatory supplemental oxygen.
16. Known additional malignancy that is progressing or has required active treatment within the past 2 years.
17. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ, excluding carcinoma in situ of the bladder, that have undergone potentially curative therapy are not excluded. Participants with low-risk early-stage prostate cancer (T1-T2a, Gleason score ≤6, and PSA <10 ng/mL) either treated with definitive intent or untreated in active surveillance with stable disease are not excluded.
18. Known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable (ie, without evidence of progression) for at least 4 weeks as confirmed by repeat imaging performed during the study screening, are clinically stable and have not required steroid treatment for at least 14 days before the first dose of study intervention.
19. Active autoimmune disease that has required systemic treatment in past 2 years except replacement therapy (eg, thyroxine or physiologic corticosteroid).
20. History of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
21. Any active bacterial, viral, or fungal infection requiring systemic therapy.
22. History or current evidence of any condition, therapy, laboratory abnormality, or other circumstance that might confound the results of the study or interfere with the participant's ability to cooperate with the requirements of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.
23. Severe hypersensitivity (≥Grade 3) to FX-909 and pembrolizumab and/or any of its excipients.

    Other Exclusions
24. History of stem cell/solid organ transplant.
25. Participants who have not adequately recovered from major surgery or have ongoing surgical complications.
26. Need or anticipated need for treatment with a prohibited therapy described in Section 21.11.2 during the treatment phase of this study
27. If female, is pregnant, breastfeeding, or expecting to conceive, or if male, expect to father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study drug.
28. Participant is or has an immediate family member who is a member of the study site or Sponsor staff directly involved with this study, unless prospective IRB or EC approval is given allowing exception to this criterion.
29. Participants with any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
30. Any condition that, in the opinion of the Investigator, would interfere with evaluation of the investigational product or interpretation of the participant's safety or study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-08-24 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
To assess dose-limiting toxicities, the incidence and severity of adverse events and serious adverse events associated with FX-909 (Safety and Tolerability) | through study completion, an average of 3 years
  Incidence of dose-limiting toxicities (DLTs); Incidence and severity of adverse events (AEs) and serious adverse events (SAEs)

SECONDARY OUTCOMES:
To define the preliminary recommended phase 2 dose of FX-909, and/or maximum tolerated dose (MTD) | through study completion, an average of 3 years
  Assess patients' safety measures (AEs/SAEs) in comparison with patients' objective response rates
To characterize the pharmacokinetic profile of FX-909 in patients with advanced solid malignancies | through study completion, an average of 3 years
  Plasma pharmacokinetic parameters of FX-909 via AUC
To characterize the pharmacokinetic profile of FX 909 in patients with advanced solid malignancies | through study completion, an average of 3 years
  Plasma pharmacokinetic parameters of FX-909, via Cmax
To characterize the pharmacokinetic profile of FX 909 in patients with advanced solid malignancies | through study completion, an average of 3 years
  Plasma pharmacokinetic parameters of FX-909, via Tmax
To characterize the pharmacokinetic profile of FX 909 in patients with advanced solid malignancies | through study completion, an average of 3 years
  Plasma pharmacokinetic parameters of FX-909 via T½
To characterize the pharmacokinetic profile of FX 909 in patients with advanced solid malignancies | through study completion, an average of 3 years
  Plasma pharmacokinetic parameters of FX-909 via renal clearance in urine
To characterize the pharmacokinetic profile of FX 909 in patients with advanced solid malignancies | through study completion, an average of 3 years
  Plasma pharmacokinetic parameters of FX-909 via percentage of FX-909 in urine
To evaluate preliminary antitumor activity of FX 909 in patients with advanced solid malignancies | through study completion, an average of 3 years
  Objective response rate (ORR)
To evaluate preliminary antitumor activity of FX 909 in patients with advanced solid malignancies | through study completion, an average of 3 years
  Duration of Response (DoR)
To evaluate preliminary antitumor activity of FX 909 in patients with advanced solid malignancies | through study completion, an average of 3 years
  Time to response
To evaluate preliminary antitumor activity of FX 909 in patients with advanced solid malignancies | through study completion, an average of 3 years
  Disease Control Rate (DCR)
To evaluate preliminary antitumor activity of FX 909 in patients with advanced solid malignancies | through study completion, an average of 3 years
  Progression-Free Survival (PFS) based on Investigator assessment using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria
To evaluate preliminary antitumor activity of FX 909 in patients with advanced solid malignancies | through study completion, an average of 3 years
  Overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Gopa Iyer, MD, Principal Investigator — Memorial Slone Kettering
Locations (11):
- United States (11):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Yale Cancer Center, New Haven, Connecticut
  - The University of Chicago Medicine, Chicago, Illinois
  - Mass General Cancer Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Memorial Slone Kettering Cancer Center, New York, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Houston Methodist Cockrell Center for Advanced Therapeutics, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
study data
Supporting Information: Study Protocol, ICF, CSR